CLINICAL TRIAL: NCT03310645
Title: Two-part, Double-blind, Placebo-controlled, Randomized, Parallel-group Study: (Part 1) in Healthy Male Volunteers to Assess Safety and Tolerability of Ascending Repeated Oral Doses of BAY1817080, Followed by (Part 2), Two-way Crossover Administration of Four Different Doses in Patients With Refractory Chronic Cough to Assess Safety, Tolerability and Efficacy for Proof of Concept
Brief Title: Repeat Doses of BAY 1817080 in Healthy Males & Proof of Concept in Chronic Cough Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18184; 2017-001620-22 (EudraCT Number)
Record Dates: First submitted 2017-09-28; First posted 2017-10-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cough
Keywords: Refractory chronic cough; healthy volunteers
MeSH Terms: conditions — Cough; Chronic Cough

STUDY DESIGN:
Intervention Model Description: Part 1: Ascending multiple doses in healthy volunteers Part 2: Ascending doses within two-way crossover design in patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose 1 of BAY1817080 (Experimental): Study Part 1:
  Oral dose 1 of BAY1817080 twice daily with a loading dose administered three times on Day 1
  Interventions: Drug: BAY1817080
- Dose 2 of BAY1817080 (Experimental): Study Part 1:
  Oral dose 2 of BAY1817080 twice daily with a loading dose administered three times on Day 1
  Interventions: Drug: BAY1817080
- Dose 3 of BAY1817080 (Experimental): Study Part 1:
  Oral dose 3 of BAY1817080 twice daily with a loading dose administered three times on Day 1
  Interventions: Drug: BAY1817080
- Dose 4 of BAY1817080 (Experimental): Study Part 1:
  Oral dose 4 of BAY1817080 twice daily with a loading dose administered three times on Day 1
  Interventions: Drug: BAY1817080
- Placebo (Placebo Comparator): Study Part 1:
  Oral dose of matching placebo twice daily with a loading dose administered three times on Day 1
  Interventions: Drug: Matching Placebo
- Placebo+BAY1817080 (Experimental): Study Part 2:
  Randomized crossover design in cough patients Placebo+4 different doses of BAY1817080
  Interventions: Drug: BAY1817080; Drug: Matching Placebo
- BAY1817080+Placebo (Experimental): Study Part 2:
  Randomized crossover design in cough patients 4 different doses of BAY1817080+Placebo
  Interventions: Drug: BAY1817080; Drug: Matching Placebo

INTERVENTIONS:
Drug: BAY1817080 — 4 different doses over the course of study
  Arms: BAY1817080+Placebo; Dose 1 of BAY1817080; Dose 2 of BAY1817080; Dose 3 of BAY1817080; Dose 4 of BAY1817080; Placebo+BAY1817080
Drug: Matching Placebo — Matching placebo for BAY1817080
  Arms: BAY1817080+Placebo; Placebo; Placebo+BAY1817080

SUMMARY:
To investigate the safety and tolerability of ascending repeated oral doses of BAY1817080 in healthy volunteers(Part1).

To investigate the safety, tolerability and efficacy of BAY1817080 in patients with refractory chronic cough(Part2).

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Male; healthy according to complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12 lead ECG, clinical laboratory tests
* Age: 18-45 years (inclusive) at the first screening visit.
* Non-smoker for at least the past 6 months and with a pack year history of equal to or less than 5 years.
* Subjects who are sexually active and have not been surgically sterilized must agree to use two reliable and acceptable methods of contraception simultaneously when having sexual intercourse with women of childbearing potential (one method used by the subject and one method used by the partner) during the study and for 90 days after receiving the investigational medicinal product and not to act as sperm donor for 90 days after dosing. [Acceptable methods of contraception include for example: (a) condoms (male or female) with or without a spermicidal agent, (b) diaphragm or cervical cap with spermicide, (c) intrauterine device, (d) hormone-based contraception.

Part 2:

* Age: >18 years at the first screening visit
* Refractory chronic cough for at least one year:

  * that has been shown to be unresponsive to at least 8 weeks of targeted treatment for identified underlying triggers including reflux disease, asthma and post-nasal drip or unexplained cough, and
  * for which no objective evidence of an underlying trigger can be determined after investigation.
* Score of >40 mm on the Cough Severity visual analogue scale (VAS) at screening.
* For male patients:

Male patients who are sexually active and have not been surgically sterilized must agree to use two reliable and acceptable methods of contraception simultaneously (one method used by the study patient and one method used by the partner) during the study and for 90 days after receiving the investigational medicinal product and not to act as sperm donor for 90 days after dosing. [Acceptable methods of contraception include for example: (a) condoms (male or female) with or without a spermicidal agent, (b) diaphragm or cervical cap with spermicide, (c) intrauterine device, (d) hormone-based contraception.

--For female patients: Confirmed post-menopausal woman (defined as exhibiting spontaneous amenorrhea for at least 12 months before screening or as exhibiting spontaneous amenorrhea for 6 months before screening with documented serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL) or Woman without childbearing potential based on surgical treatment at least 6 weeks before screening such as bilateral tubal ligation, bilateral oophorectomy with or without hysterectomy (documented by medical report verification) or Woman of childbearing potential that agrees to use two reliable and acceptable methods of contraception simultaneously (one method used by the study patient and one method used by the partner) during the study and for at least 10 days after the last dose. Acceptable methods of contraception include for example: (a)condoms (male or female) with or without a spermicidal agent (b)diaphragm or cervical cap with spermicide (c) intrauterine device (d)hormone-based contraception.

Exclusion Criteria:

Part 1

* Relevant diseases potentially interfering with the study's aims (e.g.respiratory diseases) within the four weeks before screening or between screening and randomization
* Any febrile illness within the four weeks before screening or between screening and randomization
* Medical history of hypogeusia/dysgeusia or the subject has a dysfunction in his/her ability to taste, as revealed by the taste disturbance questionnaire during screening and the pre dose procedures
* Use of any over-the-counter cough mixture within the 24 hours before screening

Part 2:

* FEV1 or FVC of less than 60% of predicted normal, at screening
* History of upper or lower respiratory tract infection or recent significant change in pulmonary status within the 4 weeks before baseline visit.
* Current smoking habit or history of smoking within the 6 months before the screening visit.
* History of smoking (at any time) for more than 20 pack-years in total (20 cigarettes per pack)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events in study part 1 | Up to 5 weeks
Severity of treatment emergent adverse events in study 1 | Up to 5 weeks
  The intensity of an AE is classified according to the following categories:
  * Mild: A type of adverse event that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living.
  * Moderate: A type of adverse event that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant.
  * Severe: A type of adverse event that requires intensive therapeutic intervention. The event interrupts usual activities of daily living, or significantly affects clinical status
Frequency of treatment emergent adverse events in study part 2 | Up to 12 weeks
Severity of treatment emergent adverse events in study part 2 | Up to 12 weeks
  The intensity of an AE is classified according to the following categories:
  * Mild: A type of adverse event that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living.
  * Moderate: A type of adverse event that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant.
  * Severe: A type of adverse event that requires intensive therapeutic intervention. The event interrupts usual activities of daily living, or significantly affects clinical status
24-hour cough counts | At week 1 in period A
24 hour cough counts | At week 2 in period A
24 hour cough counts | At week 3 in period A
24 hour cough counts | At week 1 in period B
24 hour cough counts | At week 2 in period B
24 hour cough counts | At week 3 in period B

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United Kingdom (7):
  - North Tyneside General Hospital, North Shields, Tyne and Wear
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Queen's University, Belfast
  - Castle Hill Hospital, Cottingham
  - King's College Hospital - NHS Foundation Trust, London
  - University Hospital of South Manchester, Manchester
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Reif S, Schultze-Mosgau MH, Engelen A, Piel I, Denner K, Roffel A, Tiessen R, Klein S, Francke K, Rottmann A. Mass Balance and Metabolic Pathways of Eliapixant, a P2X3 Receptor Antagonist, in Healthy Male Volunteers. Eur J Drug Metab Pharmacokinet. 2024 Jan;49(1):71-85. doi: 10.1007/s13318-023-00866-0. Epub 2023 Dec 3. PMID 38044419
- [Derived] Friedrich C, Francke K, Gashaw I, Scheerans C, Klein S, Fels L, Smith JA, Hummel T, Morice A. Safety, Pharmacodynamics, and Pharmacokinetics of P2X3 Receptor Antagonist Eliapixant (BAY 1817080) in Healthy Subjects: Double-Blind Randomized Study. Clin Pharmacokinet. 2022 Aug;61(8):1143-1156. doi: 10.1007/s40262-022-01126-1. Epub 2022 May 28. PMID 35624408
- [Derived] Morice A, Smith JA, McGarvey L, Birring SS, Parker SM, Turner A, Hummel T, Gashaw I, Fels L, Klein S, Francke K, Friedrich C. Eliapixant (BAY 1817080), a P2X3 receptor antagonist, in refractory chronic cough: a randomised, placebo-controlled, crossover phase 2a study. Eur Respir J. 2021 Nov 18;58(5):2004240. doi: 10.1183/13993003.04240-2020. Print 2021 Nov. PMID 33986030
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/